CLINICAL TRIAL: NCT06077838
Title: A Single-Center Phase 3 Study of RELAXaHEAD: A Behavioral Approach to Remote Migraine Management in Primary Care
Brief Title: RELAXaHEAD for Headache Patients (Phase III)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-01208
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Migraine
Keywords: Migraine; Smartphone App; Headache Diary; Headache Tracking
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RELAX Group 1 (Active Comparator): Participants will receive access to the RELAXaHEAD app version 1 which contains certain features for migraine self-management with written materials.
  Interventions: Behavioral: RELAXaHEAD Smartphone App Version 1
- RELAX Group 2 (Active Comparator): Participants will receive access to the RELAXaHEAD app version 2 which contains certain features for migraine self-management with written and audio materials.
  Interventions: Behavioral: RELAXaHEAD Smartphone App Version 2

INTERVENTIONS:
Behavioral: RELAXaHEAD Smartphone App Version 1 — RELAXaHEAD is a smartphone application that allows users to track headache frequency and severity, sleep, medication, medication side effects, and menstrual cycle, and create personal notes daily. The RELAXaHEAD app has an option for users to view their data reports and charts.
  Arms: RELAX Group 1
Behavioral: RELAXaHEAD Smartphone App Version 2 — RELAXaHEAD is a smartphone application that allows users to track headache frequency and severity, sleep, medication, medication side effects, and menstrual cycle, and create personal notes daily. The RELAXaHEAD app has an option for users to view their data reports and charts. This version also contains audio materials.
  Arms: RELAX Group 2

SUMMARY:
This study is a fully powered, remote randomized control trial to evaluate RELAXaHEAD in people with migraine.

DETAILED DESCRIPTION:
Patients with migraine seen across diverse primary care practices (through three different affiliated hospitals and one of the largest family health center groups in the country) will be identified via an electronic medical record system. The investigators will randomize 356 participants and examine the potential benefits to two different smartphone based interventions between baseline and weeks 3-6. The investigators will also examine the persistence of effects up to 26 weeks post-treatment, mediators to explore mechanisms, and moderators to identify subgroups of patients for whom the intervention seems most effective.

ELIGIBILITY:
Inclusion Criteria:

* English speaking. (At this time, the validated app is only available in English.)
* ≥16 years of age
* Meets International Classification of Headache Disorder (ICHD)-3 migraine criteria based on Information in the Study Manual
* Headaches for ≥1 year with a stable pattern for the past >3 months
* Agreement to not make any preventive medication changes for the 3 months before the start of the trial and then the 6 weeks of the intervention part of the study
* 4-29 headache days a month (so that we include those in whom we typically offer preventive treatment (>4 headache days/month and those with more frequent migraines including chronic migraine but exclude those with continuous headaches (30 days/month))
* MSQv2 score <75 for role restrictive function to ensure participants have sufficient reduced quality of life to potentially benefit from the intervention (see if there is a positive effect of the intervention)

Exclusion Criteria:

* Patients who have had CBT, Biofeedback, or other Relaxation Therapy for migraine in the past year
* Alcohol or other substance abuse as determined by self-report or prior documentation in the medical record
* Diagnosis of medication overuse headache and/or opioid or barbiturate use
* PHQ-8 scores greater than 15, indicate a conservative score of moderately severe depressive symptoms based on the PHQ-9 12-14 (in those with PHQ-8 scores >15, more intense intervention targeted to the depression may be needed, as depression is a significant predictor of migraine chronification and people with migraine and comorbid depression are more likely to be refractory to migraine treatments and to suffer from medication overuse)
* Unable or unwilling to follow a treatment program that relies on written and audio-taped materials
* Not having a smartphone (we do not believe this exclusion criterion will adversely affect equitable subject selection because the subject population specific to our research question would only be able to access this application via smartphone if it were to become publicly available, including subjects without smartphones would not be pertinent to our research question and overall study goals).
* Pregnant (because hormonal fluctuations in pregnancy can affect migraine outcomes)

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Modified Monthly Migraine Disability Assessment Scale (mMIDAS) Score | Baseline, Week 6
  5-item scale designed to measure disability over the previous 4 weeks. The total score is the sum of missed days due to a migraine from paid work, school, housework, and nonwork (family, social, and leisure) activities and days at paid work or housework where productivity was reduced by at least half. A decrease in scores indicates disability decreased during the observational period.

SECONDARY OUTCOMES:
Change in Migraine Specific Quality of Life (MSQ) Version 2 Scores | Baseline, Week 6
  14-item self-assessment of how migraine affects a patient's life. Items ranked on a 6-point Likert scale, where: 1 = None of the time; 2 = A little bit of the time; 3 = Some of the time; 4 = A good bit of the time; 5 = Most of the time; and 6 = All of the time. Raw dimension scores are computed as a sum of item responses and rescaled on a 0-100 scale; higher scores indicate better quality of life.
Change in Monthly Headache Days (MHDs) | Baseline, Week 6
  MHDs data derived from the mMIDAS questionnaire and electronic diary.

CONTACTS AND LOCATIONS:
Overall Officials: Mia T Minen, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: mia.minen@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to mia.minen@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.